CLINICAL TRIAL: NCT00599807
Title: Role of Vitamin D in Secondary Prevention of Knee Osteoarthritis: A Double-blind Randomized Controlled Trial
Brief Title: Zurich Multiple Endpoint Vitamin D Trial in Knee OA Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Tufts University (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PP00B-114864; 2007DR4347 (Other: Swiss Agency for Therapeutic Products (Swissmedic))
Record Dates: First submitted 2008-01-10; First posted 2008-01-24 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: 2000 IU D3/day (Active Comparator): 2000 IU vitamin D3 taken orally each day for 2 years
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- 2: 800 IU D3 / day (Active Comparator): 800 IU vitamin D3 taken orally each day for 2 years
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — the intervention is a dietary supplement comparing the current standard (800 IU) to the current safe upper limit (2000 IU)

SUMMARY:
This is a 2-year double-blind randomized controlled trial in 287 community-dwelling individuals age 60 years or older undergoing uni-lateral total knee replacement due to severe OA of the knee.We compare an oral dose of 2000 IU vitamin D3 per day to 800 IU. The primary endpoints are pain and disability related to rehabilitation of the operated knee,and related to the expected high prevalence of OA in the contra-lateral knee. Secondary endpoints are change in 25(OH)D levels, muscle strength, balance, lower extremity function, the rate of falls, bone density and bone quality, bone metabolism, general pain, fall-related fractures, body composition, blood-pressure, major cardiovascular events, blood glucose-insulin levels, executive cognitive function, rate of upper respiratory tract infections / all infections, tooth loss, dental health, health care utilization, number and size of facial skin keratosis, and radiographic progression of the non-operated knee. Pain and disability will be assessed by the pain and function subscales of the Western Ontario- McMaster Universities Osteoarthritis Index (WOMAC). Randomization will be stratified by WOMAC function prior to surgery, radiological evidence for OA in the contra-lateral knee, and hospital. Clinical visits will take place at baseline (6-8 weeks after TKR), at 6, 12, 18 and 24 months of treatment. In addition, all individuals will receive a phone call every 2 month to assess adverse outcomes and compliance to treatment, supported by a hotline for immediate report of adverse events.

Statistical power: We expect more than 80% power with 200 participants completing their 24 month follow-up, and 260 participants completing their 12 month follow-up.

This is a trial with medicinal product.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral knee replacement due to knee osteoarthritis
* Age 60+ years
* German language skills
* community dwelling

Exclusion Criteria:

* Bi-lateral knee replacement or hip replacement planned in the trial period, or in the previous 6 months
* Chronic steroid intake
* Serum calcium corrected for serum albumin > 2.6 mmol/l
* GFR < 30 ml/min
* Severe visual or hearing impairment
* Inflammatory arthritis
* Malabsorption
* High alcohol intake
* Sarcoidosis, primary hyperparathyroidism
* History of kidney stones, lymphoma
* Chemotherapy for cancer in the previous 12 months
* Hemiplegia
* Morbus Parkinson
* Unable to walk 3 meters prior to surgery
* Bisphosphonate, parathyroid hormone , fluoride or calcitonine therapy in the last 6 months
* Zolendronate in the last year
* M. Paget (Ostitis deformans)
* Vitamin D3 intake more than 800IU/d over more than 1 month
* stay on a sunny location for more than 6 weeks per year
* heart failure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2008-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
pain and function of the operated and non-operated knee | 0, 6,12,18, 24 months
rate of falls | 0, 24 months

SECONDARY OUTCOMES:
strength, balance, function, physical activity | 0,6,12,18,24 months
bone density, bone quality | 0, 24 months
body composition | 0, 24 months
blood pressure | 0,12,24 months
number of teeth | 0, 24 months
cost, health care utilization | 0,6,12,18,24 months
facial skin keratosis (number and size) | 0, 24 months
cognitive function | 0, 24 months
depression, mental health | 0,12,24 months
fasting blood glucose - insulin levels | 0,12,24
Number of upper respiratory infections and number of any infections | 0, 6,12,28,24
bone metabolism | 0,6,12,18,24
radiographic progression of the non-operated knee | 0, 24 months
general pain | 0,6,12,18,24 months
Quality of life | 0,6,12,18,24

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, MD, MPH, Principal Investigator — University Hospital Zurich, Centre on Aging and Mobility
Locations (1):
- University Hospital Zurich, Centre on Aging and Mobility, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Braendle K, Egli A, Bischoff-Ferrari H, Freystaetter G. Does living alone influence fall risk among Swiss older adults aged 60+? A pooled observational analysis of three RCTs on fall prevention. BMJ Open. 2024 May 20;14(5):e081413. doi: 10.1136/bmjopen-2023-081413. PMID 38772577
- [Derived] Abderhalden LA, Meyer S, Dawson-Hughes B, Orav EJ, Meyer U, de Godoi Rezende Costa Molino C, Theiler R, Stahelin HB, Ruschitzka F, Egli A, Forman JP, Willett WC, Bischoff-Ferrari HA. Effect of daily 2000 IU versus 800 IU vitamin D on blood pressure among adults age 60 years and older: a randomized clinical trial. Am J Clin Nutr. 2020 Sep 1;112(3):527-537. doi: 10.1093/ajcn/nqaa145. PMID 32542307
- [Derived] Freystaetter G, Fischer K, Orav EJ, Egli A, Theiler R, Munzer T, Felson DT, Bischoff-Ferrari HA. Total Serum Testosterone and Western Ontario and McMaster Universities Osteoarthritis Index Pain and Function Among Older Men and Women With Severe Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2020 Nov;72(11):1511-1518. doi: 10.1002/acr.24074. PMID 31557423
- [Derived] Schietzel S, Fischer K, Brugger P, Orav EJ, Renerts K, Gagesch M, Freystaetter G, Stahelin HB, Egli A, Bischoff-Ferrari HA. Effect of 2000 IU compared with 800 IU vitamin D on cognitive performance among adults age 60 years and older: a randomized controlled trial. Am J Clin Nutr. 2019 Jul 1;110(1):246-253. doi: 10.1093/ajcn/nqz081. PMID 31152541